CLINICAL TRIAL: NCT01831245
Title: Right-sided Colon Tumor, Laparoscopic and Open Surgery, in an ERAS Protocol
Brief Title: Right-sided Colon Tumor, Laparoscopic Versus Open Surgery, in an ERAS Protocol
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Region Örebro County (Other); Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Ulf Gustafsson, MD, PhD, Karolinska Institutet
Other Study IDs: 2012/2105-31/2
Record Dates: First submitted 2013-02-25; First posted 2013-04-15 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Colon Tumor
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Register study. Patients who had been operated for right-sided colon tumor or benign adenoids between year 2011 to 2012. The study compare open surgery with laparoscopic surgery in an ERAS (Enhanced Recovery After Surgery) protocol.

Hypothesis:

Operation of right-sided colon tumor and large benign adenoids, a better selection of patients for open or laparoscopic surgery can improve short term results.

ELIGIBILITY:
Inclusion Criteria:

* right-sided colon tumor or large benign adenoids

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Right sided colom tumor or large benign adenoids
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pathological Anatomic diagnosis (PAD) on a tumor biopsy | day of surgery
  After PAD result, malign or benign tumor, type of malign tumor,tumor growth, stage, lymphatic recharge.
  Right selection of patients to laparoscopic versus open surgery in relation to PAD result?

SECONDARY OUTCOMES:
Length of hospital stay, days | 30 days after surgery
  Compare laparoscopic versus open surgery
C - reactive protein | 1-7 days after surgery
  Inflammation answer laparoscopic versus open surgery

OTHER OUTCOMES:
Immobilizing patient after surgery | 4 -10 hours after surgery
  After laparoscopic versus open surgery
Leakage of anastomosis | 0 - 30 days after surgery
  Compare laparoscopic versus open surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Gustafsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Örebro University Hospital, Örebro
  - Ersta Hospital, Stockholm
  - Danderyds Hospital, Stockholm